CLINICAL TRIAL: NCT02432352
Title: Our Family Our Future: Family Prevention of HIV Risk and Depression in HIV-endemic South Africa
Brief Title: Our Family Our Future: Acceptability and Feasibility Study of a Family Prevention Program for HIV Risk and Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Caroline Kuo, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K01MH096646 (NIH)
Record Dates: First submitted 2015-04-19; First posted 2015-05-04 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Sexual Behavior; Depression
MeSH Terms: conditions — Sexual Behavior; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Families are randomly allocated to a behavioral intervention arm (called Our Family Our Future) focusing on reducing sexual risk behavior in adolescents and reducing or maintaining symptoms that fall below the clinically significant range for depression. Arms will be allocated using urn randomization.
  Interventions: Behavioral: Our Family Our Future
- Control (No Intervention): Families are randomly allocated to the control arm (which receives standard usual care, and then offered the intervention after outcome assessments as a wait-list) using urn randomization.

INTERVENTIONS:
Behavioral: Our Family Our Future — The Our Family Our Future Program is a family preventive intervention that uses resilience and prevention focused strategies to reduce sexual risk behaviors and build mental wellbeing among adolescents.
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of a family-based preventive intervention designed to reduce sexual risk behaviors and depressive symptoms among South African adolescents and their parents/guardians/caregivers.

DETAILED DESCRIPTION:
The Our Family Our Future Program is a preventive intervention program designed to prevent or reduce adolescent sexual risk behavior and to increase mental health resilience against depression onset among adolescents (13-15 years of age). The intervention takes a family approach and addresses HIV risk and depression in an integrated model. HIV and depression are the leading causes of global burden of disease in low and middle income countries. The intervention is being tested in South Africa, the country confronting the largest HIV epidemic in the world and because preliminary studies with South African families identified poor mental health and sexual risk behavior as priority areas for preventive intervention development and testing.

This study is a randomized pilot design, where 152 adolescents and parents will be randomly assigned to an intervention condition or a standard usual care condition and then offered the experimental intervention as on a wait-list. Families will be recruited and screened for eligibility based on systematic house-to-house recruitment in the community. Eligibility is based on dyadic eligibility and includes age criteria, consistent presence in the household, depressive symptoms that fall below clinically significant threshold criteria, and ability to provide informed consent and assent. Eligible families will be randomized and offered a preventive intervention program in a group format, led by program facilitators in a community setting. The intervention program consists of 3 sessions plus an individualized family meeting. In some modules parents/guardians/caregivers and adolescents will have content delivered together and in some modules parents/guardians/caregivers and adolescents will break out to adult-only or adolescent-only groups.

The overall objective of study is to assess the following study questions:

Question 1: Is this study feasible? Question 2: Is this intervention acceptable to the target population? Question 3: Is there preliminary evidence of hypothesized effects of the intervention, that the intervention will reduce or maintaining symptoms that fall below the clinically significant range for depression and reduce or delay actual or intended sexual risk behavior in adolescents?

The study takes a single blind, randomized pilot trial. The study takes a secondary prevention approach. The investigators collect three sets of data. First, the investigators assess feasibility by examining recruitment rates, attendance, completion, and drop-out rates, and fidelity. Second, the investigators assess acceptability by examining satisfaction data. Third, as a secondary aim, the investigators use pilot data to assess hypothesized intervention effects by examining outcomes at baseline, immediately post-intervention (2-4 weeks after the last intervention session is completed), and at four months.

ELIGIBILITY:
Inclusion Criteria:

PARENTS/GUARDIANS/CAREGIVERS

1. 18+ years
2. primary caregiver or the person responsible for childcare in the household on a day to day basis (as identified by the household);
3. when more than one primary caregiver exists in the household, one will be chosen at random;
4. lives in the household at least 4 days a week
5. sub clinical thresholds of depressive symptoms

Adolescent inclusion criteria are:

1. 13-15 years;
2. concurs that the adult identified is their primary caregiver;
3. when more than one child in the family falls within the eligible age range, one child will be chosen at random;
4. lives in the household at least 4 days a week;
5. sub clinical thresholds of depressive symptoms

Exclusion Criteria:

PARENTS/GUARDIANS/CAREGIVERS & Adolescents

1. cognitive impairments that would not allow them to provide informed consent or assent;
2. if they participated in qualitative phases of the study
3. report no or low symptoms or clinically significant thresholds of depression -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sexual behavior or intended sexual behavior at 4 months post-intervention | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
  as measured through lifetime and past 3 month sexual acts, condom use, HIV and STI status, prior pregnancy
Change or maintenance of depressive symptoms at sub-clinical range from baseline to 4 months post-intervention measured by CES-D and CES-DC | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
  Self-reported depressive symptoms
Intervention acceptability - satisfaction with intervention content, delivery, length using the client satisfaction questionnaire and as measured on a likert scale response and as open-ended response options | acceptability will be assessed during the intervention, an expected average timeframe of 4 weeks
Intervention feasibility measured by attendance, retention for outcome assessments, fidelity | cceptability will be assessed during the intervention, an expected average timeframe of 4 weeks

SECONDARY OUTCOMES:
Change in resilience from baseline to 4 months post-intervention as measured through CD-RISC | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in depression impairment from baseline to 4 months post-intervention as measured through DISP and CPODMV | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in perceived HIV risk susceptibility from baseline to 4 months post-intervention using a ranking derived from a 0-100 and as measured on a likert scale response | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in HIV knowledge from baseline to 4 months post-intervention as measured through the HIV Knowledge Questionnaire | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in HIV stigma from baseline to 4 months post-intervention as measured through the HIV Knowledge Questionnaire | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in norms and attitudes about sex from baseline to 4 months post-intervention as measured on a likert scale response | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in norms and attitudes about condoms from baseline to 4 months post-intervention as measured through the condom attitudes scale and likert response questions | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in sexual behavior self-efficacy from baseline to 4 months post-interventionusing a ranking derived from a 0-100 and as measured on a likert scale response | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in anxiety from baseline to 4 months post-interventionas measured through BAI and RCMAS | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in psychological distress from baseline to 4 months post-intervention as measured through K6 and SDQ | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in trauma symptoms from baseline to 4 months post-intervention as measured through PCL and NSESSS | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in substance use from baseline to 4 months post-intervention as measured through AUDIT and DUDIT | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in hope from baseline to 4 months post-intervention as measured through BHS | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in social support from baseline to 4 months post-intervention as measured through MSPSS | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in family relationship from baseline to 4 months post-intervention as measured through Family Relationship Scale | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in family communication from baseline to 4 months post-intervention as measured through the Parent-adolescent Communication Scale | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in family communication from baseline to 4 months post-intervention as measured through the Parent-adolescent Sex Communication Scale | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in family relationship from baseline to 4 months post-intervention as measured through the Inventory of Parent-peer Attachment | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in parenting from baseline to 4 months post-interventionas measured through the Parental Monitoring Questionnaire | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention
Change in parenting from baseline to 4 months post-intervention as measured through the Parenting Scale | assessed at baseline, starting within 2-4 weeks of intervention end, and 4 months post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Caroline Kuo, Cape Town, Western Cape, South Africa

REFERENCES:
- [Result] Kuo C, Atujuna M, Mathews C, Stein DJ, Hoare J, Beardslee W, Operario D, Cluver L, K Brown L. Developing family interventions for adolescent HIV prevention in South Africa. AIDS Care. 2016;28 Suppl 1(sup1):106-10. doi: 10.1080/09540121.2016.1146396. Epub 2016 Feb 26. PMID 26916841
- [Result] Kuo C, LoVette A, Stein DJ, Cluver LD, Brown LK, Atujuna M, Gladstone TRG, Martin J, Beardslee W. Building resilient families: Developing family interventions for preventing adolescent depression and HIV in low resource settings. Transcult Psychiatry. 2019 Feb;56(1):187-212. doi: 10.1177/1363461518799510. Epub 2018 Oct 5. PMID 30289374
- [Result] Kuo C, Mathews C, LoVette A, Harrison A, Orchowski L, Pellowski JA, Atujuna M, Stein DJ, Brown LK. Perpetration of sexual aggression among adolescents in South Africa. J Adolesc. 2019 Apr;72:32-36. doi: 10.1016/j.adolescence.2019.02.002. Epub 2019 Feb 13. PMID 30771665
- [Result] Kuo C, LoVette A, Pellowski J, Harrison A, Mathews C, Operario D, Beardslee W, Stein DJ, Brown L. Resilience and psychosocial outcomes among South African adolescents affected by HIV. AIDS. 2019 Jun 1;33 Suppl 1(Suppl 1):S29-S34. doi: 10.1097/QAD.0000000000002177. PMID 31397720
- [Result] Kuo C, Mathews C, Giovenco D, Atujuna M, Beardslee W, Hoare J, Stein DJ, Brown LK. Acceptability, Feasibility, and Preliminary Efficacy of a Resilience-Oriented Family Intervention to Prevent Adolescent HIV and Depression: A Pilot Randomized Controlled Trial. AIDS Educ Prev. 2020 Feb;32(1):67-81. doi: 10.1521/aeap.2020.32.1.67. PMID 32202920